CLINICAL TRIAL: NCT03559218
Title: Pilot Study: KeraStat(R) Cream for Radiation Dermatitis
Brief Title: KeraStat(R) Cream for Radiation Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KeraNetics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSCM-CRD-001
Record Dates: First submitted 2018-03-19; First posted 2018-06-18 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Standard of care (Other): Patients undergoing radiation therapy for breast cancer will be provided instructions for radiation dermatitis per institutional standard of care
  Interventions: Other: Standard of care
- KeraStat Cream (Experimental): Patients undergoing radiation therapy for breast cancer will be provided KeraStat Cream for twice daily application.
  Interventions: Device: KeraStat(R) Cream

INTERVENTIONS:
Device: KeraStat(R) Cream — KeraStat Cream is a cream wound dressing that contains 5% keratin.
  Arms: KeraStat Cream
Other: Standard of care — Patients will be instructed to follow institutional standard of care for radiation dermatitis
  Arms: Standard of care

SUMMARY:
The primary objectives of the proposed research are to evaluate patient use of KeraStat Cream and collect data to inform a larger future trial.

DETAILED DESCRIPTION:
The primary objectives of the proposed research are to evaluate patient use of KeraStat Cream and collect data to inform a larger future trial.

The secondary objectives are to assess the safety and tolerability of KeraStat Cream in subjects at risk of radiation dermatitis, to assess the effectiveness of KeraStat Cream and how that compares to the current standard of care, and to estimate the amount of KeraStat Cream used per patient and coverage on skin.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70
2. Female
3. Diagnosis of breast cancer and scheduled to receive 4 to 6 weeks of radiation therapy (radiation dose of 42 Gy or more)
4. Able and willing to sign protocol consent form
5. Able and willing to document symptoms and treatment details as often as needed, not to exceed daily notes
6. Able and willing to have photographs of the affected area taken regularly

Exclusion Criteria:

1. Women who are pregnant, lactating/nursing or plan to become pregnant
2. Previous radiation therapy to the area to be treated with radiation therapy
3. Receiving palliative radiation therapy
4. Unhealed or infected surgical sites in the irradiation area
5. Patients undergoing cytotoxic chemotherapy or concurrent Herceptin as part of overall treatment plan (tamoxifen/aromatase inhibitor allowed)
6. Use of oral corticosteroids or topical corticosteroids in the irradiation area
7. Autoimmune disease
8. Skin disease in target irradiation area
9. Known allergy to the standard of care or ingredients in KeraStat Cream

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Winfield, MD PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care | KeraStat Cream
Started | 12 | 13
Completed | 11 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline RTOG score and DQLI score, as assessed by physician.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | KeraStat Cream | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Categorical [Count of Participants; unit: Participants] — Population: One subject withdrew at baseline prior to treatment and was not included.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 7 | 12
    >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (7.5) | 59.2 (9.9) | 62.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24
Radiation Therapy Oncology Group Skin Toxicity Grade (RTOG) [Mean (Standard Deviation); unit: units on a scale (RTOG)] — RTOG as assessed by physician: Grade 0 (no toxicity) to Grade 4 (
  Note expectation is that there would be no skin toxicity at the start of the study, so a baseline of "0" is the expected value.
  Increasing pathology is reflected in the higher grades.
  units on a scale (RTOG) | 0 (0) | 0 (0) | 0 (0)
Dermatology Life Quality Index [Mean (Standard Deviation); unit: units on a scale] — This scale measures the impact of skin conditions on a participant's quality of life. The DLQI is calculated by adding the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. A score higher than 10 indicates that the patient's life is being severely affected by their skin disease.
  units on a scale | 2.73 (5.12) | 0.31 (0.85) | 1.42 (3.89)

OUTCOME MEASURES:

1. Primary Outcome: Radiation Therapy Oncology Group Skin Toxicity Scoring
Description: The RTOG will be used to track skin reactions to radiation therapy. No toxicity is considered a 0, while massive toxicity is considered a 4. Data will be aggregated across groups at each time point.
Time Frame: Baseline (Visit 1), Weekly Visits throughout RT (Visits 2-6), Final Visit approximately 6 weeks post-RT (Visit 7). Subject study duration 8-12 weeks.
Population: One subject missed visit 5. One subject missed visit 6. Subject #18 missed visit 7.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Standard of Care | KeraStat Cream
Number analyzed (Participants) | 11 | 13
score on a scale
  Visit 1 | 0.00 [0 to 0] | 0.00 [0 to 0]
  Visit 2 | 0.09 [0 to 1] | 0.15 [0 to 1]
  Visit 3 | 0.55 [0 to 1] | 0.62 [0 to 1]
  Visit 4 | 0.82 [0 to 1] | 1.00 [0 to 2]
  Visit 5: number analyzed (Participants) | 11 | 12
  Visit 5 | 1.00 [0 to 2] | 1.17 [0 to 2]
  Visit 6: number analyzed (Participants) | 11 | 12
  Visit 6 | 1.36 [0 to 2] | 1.00 [0 to 1]
  Visit 7: number analyzed (Participants) | 10 | 13
  Visit 7 | 0.30 [0 to 1] | 0.23 [0 to 1]

2. Primary Outcome: Dermatology Life Quality Index
Description: The DLQI measures the impact of dermatological conditions on a patient's quality of life. The DLQI is scored by summing the score of each question (answered from not at all, 0, to very much, 3). The maximum is 30 and the minimum is 0. The higher the score, the greater the impairment of quality of life. Data will be aggregated across treatment groups.
Time Frame: as for outcome 1
Population: One subject missed visit 5. One subject missed visit 6. Subject #18 missed visit 7.
Measure: Mean (Full Range); unit: units on a scale (DQLI score)
Arm/Group | Standard of Care | KeraStat Cream
Number analyzed (Participants) | 11 | 13
units on a scale (DQLI score)
  Visit 1 | 2.73 [0 to 18] | 0.31 [0 to 3]
  Visit 2 | 1.64 [0 to 6] | 0.77 [0 to 5]
  Visit 3 | 1.91 [0 to 7] | 2.23 [0 to 15]
  Visit 4 | 2.36 [0 to 7] | 2.85 [0 to 11]
  Visit 5: number analyzed (Participants) | 11 | 12
  Visit 5 | 5.27 [0 to 15] | 4.75 [0 to 26]
  Visit 6: number analyzed (Participants) | 11 | 12
  Visit 6 | 6.18 [0 to 17] | 4.25 [0 to 14]
  Visit 7: number analyzed (Participants) | 10 | 13
  Visit 7 | 1.00 [0 to 6] | 0.85 [0 to 4]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Evaluate safety and tolerability of application of KeraStat Cream through comparison of adverse events reported in KeraStat Cream group versus standard of care.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | KeraStat Cream
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored throughout the course of radiation therapy (4-6 weeks) with a 4-week follow-up visit.
Description: All SAEs should be reported to the study sponsor within 24 hours of the investigator being aware of the event and reported to the IRB in accordance with IRB requirements.
Arm/Group | Standard of Care | KeraStat Cream
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03559218/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03559218/ICF_001.pdf